CLINICAL TRIAL: NCT04799418
Title: Non-Invasive Brainstem Modulation for the Treatment of Non-Motor Symptoms in Parkinson's Disease: An Open Label Extension (OLE) Study
Brief Title: STEM-PD Open Label Extension (OLE)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of efficacy.
Sponsor: Scion NeuroStim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNS-PD-003
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease; Parkinson's Disease and Parkinsonism
Keywords: Open Label Extension Study; Medical Devices; Non-Motor Symptoms (NMS); Non-Invasive Brain Stimulation; Parkinson Disease
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Intervention Model Description: All participants in this open label extension portion of the study receive active time-varying caloric vestibular stimulation treatment, however, participants were previously randomized to receive the active treatment or passive treatment in a previous randomized controlled trial.
Masking Description: Participant, care provider, investigator and outcomes assessors were all blinded to treatment allocation during the randomized controlled trial at the time of data collection in this open label extension
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- passive-active (Experimental): This group received passive treatment with the study device in a randomized controlled trial (RCT) that immediately preceded this open label extension (OLE ) trial during which participants received active (i.e., time-varying caloric vestibular stimulation ) treatment.
  Interventions: Device: Open Label Extension Study
- active-active (Experimental): This group received active (i.e., time-varying caloric vestibular stimulation) treatment with the study device in a randomized controlled trial (RCT) that immediately preceded this open label extension (OLE) trial during which participants received active treatment. Data from participants in this arm was only used for exploratory outcomes.
  Interventions: Device: Open Label Extension Study

INTERVENTIONS:
Device: Open Label Extension Study — This study will investigate the safety and efficacy of extended treatments for the management of symptoms related to PD.

SUMMARY:
This study seeks to establish the safety and efficacy of extended twice daily time-varying caloric vestibular stimulation treatments for treating symptoms associated with Parkinson's disease. Only participants who completed the STEM-PD randomized controlled trial portion (NCT04797611) are eligible to participate in the open label extension portion.

DETAILED DESCRIPTION:
Up to 220 participants will enter an open label extension study during which all study participants will receive active (i.e., time-varying caloric vestibular stimulation) treatment for 12 weeks (84 days). Study participants will be followed for 16 weeks (112 days) post treatment-cessation and then the twice daily active treatments will be re-introduced for the final 8 weeks (56 days).

ELIGIBILITY:
Inclusion Criteria:

* Completion of the study activities in the STEM-PD RCT trial (see STEM-PD RCT eligibility criteria noted below).
* Participants must be willing and able to give consent to participate in the study trial.
* Participants and investigators must expect that the participant will be able to remain on a stable regimen of concomitant therapies used for the management of PD motor and non-motor symptoms and not to introduce new medications used to treat motor or non-motor symptoms associated with PD during the first three months of the OLE (Day197).

Exclusion Criteria:

* Participant anticipates being unable to attend all visits and complete all study activities.
* Has a planned surgery scheduled to occur during the first 90 days of the OLE that would typically be followed with a prescription for pain management

STEM-PD RCT Eligibility criteria:

Inclusion:

1. Adult participants (aged 18 - 85 years inclusive).
2. Have been diagnosed with PD according to the UK Brain Bank Criteria (allowing for an exclusion in Step 2 for "more than one affected relative").
3. Participants must have demonstrated a sustained positive response to DRTs (e.g., levodopa, dopamine agonists or monoamine oxidase inhibitors) defined as either good or excellent responses (50-100%) for at least one year or moderate responses (30-49)% for at least three years prior to Screen.
4. Participant reports limitation or clinician-investigator determined limitation, based on knowledge of medical history, to one or more activities of daily living (e.g., writing, walking, bathing, dressing, eating, toileting, etc.).
5. Participants must be able and willing to consent to participate in the study for the RCT and OLE.
6. Participants must be willing and able to comply with study requirements.
7. Participants must have at minimum a moderate burden of NMS (i.e., MDS-UPDRS part Ia and part Ib summed total score ≥ 9) at study screen to avoid floor effects for the primary endpoint (MDS-NMS).
8. The principal investigator or designee must have confidence in the participant's ability to reliably use the TNM™ device, understand the assessments (provided in English only) and to complete the assessment battery within a given on-state period.
9. Must have a study partner (defined as someone who sees the participant for more than one hour a day, 3x per week) that is willing to consent and participate in the trial.
10. Participants must have capabilities to use and access smartphones for the collection of some study data and/or tablets or computers for access to telemedicine platforms.
11. Must be willing to answer questions related to sexual interest, arousal and performance in an interview with study staff.

Exclusion:

1. Women of child-bearing potential who are pregnant or plan to become pregnant during the course of the study

   • Women of child-bearing potential (i.e., are not yet either 3 years removed from their first menopausal symptom or 12 months removed from last menses), who are not abstinent or exclusively in same sex relationships must:
   * test negative for pregnancy as indicated by a negative urine pregnancy test;
   * agree to use an approved contraception method listed in section 5.3.3 for the entirety of the RCT and OLE;
2. Have a history or prior diagnosis of dementia or adjusted score ≤ 20 on the Montreal Cognitive Assessment (MoCA) at the screening visit.
3. Have experienced a myocardial infarction, angina or stroke within the past 12 months or a transient ischemic attack (TIA) within 6 months.
4. Are receiving deep brain stimulation therapy.
5. Are treated with a pump for continuous delivery of dopamine replacement therapy.
6. Have received MRI guided high intensity focused ultrasound within the past 12 months.
7. Experience frequent falls (defined as 2 or more falls in the past month related to Parkinson's disease). Parkinson's falls are defined as falls associated with bradykinesia, freezing, turning, change in posture and postural dizziness and do not include accidental falls.
8. Work night shifts.
9. Has any significant co-morbidity or illness which in the opinion of the investigator would prevent safe participation in the study, compliance with protocol requirements or which presents with symptoms that are also common in PD.
10. Demonstrate suicidality at screening (scores ≥ 4 on the C-SSRS Baseline in section "Suicidal Ideation" (In the past Month)). Participants that respond affirmatively to question 4 or 5 (In the past Month) should receive a referral for mental health counseling according to local site regulations and standards.
11. Use a hearing aid that is implanted or that cannot be easily removed and replaced.
12. Have a cochlear implant or myringotomy tubes.
13. Have chronic tinnitus that has been ongoing for at least 3 months and causes significant impairment of communication and/or impairment of activities of daily living.
14. Have previously been diagnosed with traumatic brain injury with ongoing sequela.
15. Have been diagnosed with a co-morbid neurological disorder that may present with symptoms overlapping with PD (e.g., stroke, brain tumor, epilepsy, Alzheimer's disease, multiple sclerosis, amyotrophic lateral sclerosis, atypical Parkinsonism or aneurysm).
16. Have been previously diagnosed with either clinically meaningful central vestibular dysfunction (lifetime) or have experienced clinically meaningful peripheral vestibular dysfunction within the last 12 months. For this purpose, clinically meaningful is defined as vestibular dysfunction which causes at least a minimal impairment in the individual activities of daily living (e.g., dressing, bathing, preparing food, conducting household chores, work or recreational activities).
17. In the Investigator's opinion, currently abuse alcohol, abuse drugs (including legal, illegal or prescribed drugs) or have a history of alcohol or drug dependency within the past 5 years or use any drugs excluded as noted in the Excluded Medications List
18. Have unresolved complications from a previous surgical procedure at the baseline visits, such as swelling or persistent pain, that requires medical intervention.
19. Have active ear infections, perforated tympanic membrane or labyrinthitis, as identified by a general ear examination performed by medically qualified Investigators.

29. Have a recent history of frequent ear infections (≥ 1 per year over the past two years).

21. Are currently enrolled or have participated in another interventional clinical trial within the last 30 days.

22. Have had eye surgery within the previous three months or ear surgery within the previous six months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2025-02-24 (Actual); Study Completion 2025-02-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Movement Disorder Center of Arizona, Scottsdale, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Parkinson's Disease and Movement Disorder of Boca Raton, Boca Raton, Florida
  - Headlands Research Orlando, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - University of Kansas Medical Center - Parkinson's Disease Center, Kansas City, Kansas
  - Quest Research, Farmington Hills, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - Meridian Clinical Research, Raleigh, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Veracity Neuroscience, Memphis, Tennessee
  - Houston Methodist Neurological Institute, Houston, Texas
  - Riverside Neurology Specialists, Newport News, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants (active or passive) completing NCT04797611 were eligible to enter this open label extension (OLE) study to receive active devices. NCT04797611 study was completed, however this OLE study terminated early, due to company closure. Incomplete data prevented analysis. Results posted compare the group differences by outcome measure for NCT04797611 passive participants who completed this active OLE (for passive-active only). Active-active outcomes were exploratory and so are not posted.
Groups:
- Experimental: Passive-active: This group received passive treatment with the study device in a randomized controlled trial (RCT) that immediately preceded this open label extension (OLE ) study during which participants received active (i.e., time-varying caloric vestibular stimulation) treatment.
- Experimental: Active-active: This group received active (i.e., time-varying caloric vestibular stimulation) treatment with the study device in a randomized controlled trial that immediately preceded this open label extension during which participants received active treatment. Data obtained from this group was only utilized for exploratory outcome measures.
Period: Overall Study
Arm/Group | Experimental: Passive-active | Experimental: Active-active
Started | 69 | 79
Completion of Treatment Period 1 | 66 | 76
Completion of Follow-Up Period | 47 | 57
Completed | 41 | 55
Not Completed | 28 | 24
Not completed — Death | 1 | 1
Not completed — Lack of Efficacy | 14 | 14
Not completed — Withdrawal by Subject | 10 | 7
Not completed — Adverse Event | 3 | 2

BASELINE CHARACTERISTICS:
Population: Participants in the passive-active group received passive treatment during the randomized control trial and active treatment during the open label extension. Participants in the active-active group received active treatment during both the randomized control trial and the open label extension. These two groups comprise all study participants that consented to participate in the open label extension prior to the early termination of the trial.
Groups:
- Experimental: Passive-active: This group received passive treatment with the study device in a randomized controlled trial that immediately preceded this open label extension trial during which participants received active (i.e., time-varying caloric vestibular stimulation) treatment.
- Experimental: Active-active: This group received active (i.e. time-varying caloric vestibular stimulation) treatment with the study device in a randomized controlled trial that immediately preceded this open label extension trial during which participants received active treatment. Data obtained from this group was only utilized for exploratory outcome measures.
- Total: Total of all reporting groups
Arm/Group | Experimental: Passive-active | Experimental: Active-active | Total
Number analyzed (Participants) | 69 | 79 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.8 (7.6) | 68.5 (7.5) | 68.6 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 27 | 45
  Male | 51 | 52 | 103
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 61 | 76 | 137
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Years of Education [Count of Participants; unit: Participants] — Population: This data is derived from the Montreal Cognitive Assessment, which is performed at interim visits, and not all participants that entered the OLE completed the assessment
  Participants
    > 12 Years of Education | 68 | 77 | 145
    < = 12 years of Education | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in The International Parkinson and Movement Disorder Society - Non-Motor Rating Scale (MDS-NMS) Total Score
Description: The primary endpoint is the change in MDS-NMS total score during the first treatment period during the open label extension (OLE) relative to the score at the end of the NCT04797611 randomized controlled trial (RCT) treatment period (day 113) for the passive-active treatment group compared to the change in MDS-NMS total score during the RCT treatment period relative to the pretreatment baseline. The MDS-NMS is 52-item rater-administered scale used to assess a wide range of non-motor symptoms in Parkinson's disease. It measures both frequency (0/never to 4/ >51% of the time) and severity (0/not present to 4/major distress or disturbance) of 13 domains. Each question is scored by multiplying frequency x severity. All question scores for each domain are summed, and the scores for each domain are summed to provide the Total Score (range = 0-832) with the higher score indicating greater non-motor symptom burden.
Time Frame: 3 months (NCT04797611 RCT: Day 29 - Day 113; This OLE: Day 113 to Day 197)
Population: This population received passive treatment during the RCT that preceded this phase of the study and active treatment in this OLE. Only participants who completed the assessments at least once during the pre-treatment baseline period and at both the RCT end of treatment visit and the end of treatment period 1 visit during this OLE are included in the results posted. Full data collection was not completed as the study terminated prior to collection of outcome assessments for all participants.
Measure: Mean (95% Confidence Interval); unit: change in score on a scale from baseline
Groups:
- Randomized Controlled Trial (RCT) Passive Treatment: This group received passive treatment with the study device in a randomized controlled trial that immediately preceded this open label extension during which participants received active (i.e., time-varying caloric vestibular simulation). Data is provided for change in scores after the 12 weeks of passive treatment in the randomized controlled trial.
- Open Label Extension (OLE) Active Treatment: This group received passive treatment with the study device in a randomized controlled trial that immediately preceded this open label extension during which participants received active (i.e., time-varying caloric vestibular simulation). Data is provided for change in scores after the 12 weeks of active treatment in the open label extension.
Arm/Group | Randomized Controlled Trial (RCT) Passive Treatment | Open Label Extension (OLE) Active Treatment
Number analyzed (Participants) | 64 | 64
change in score on a scale from baseline | -23.12 [-33.11 to -13.12] | 3.28 [-8.18 to 14.74]

2. Secondary Outcome: Change From Baseline in The International Parkinson and Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II
Description: The MDS-UPDRS Part II is a 13-item patient-reported assessment of activities of motor aspects of experiences of daily living. Scores range between 0-52, with the higher score indicating greater impairment to activities of daily living. This secondary endpoint evaluates the change in the MDS-UPDRS Part II score obtained during the first treatment period of this open label extension (OLE) relative to the score obtained at the end of the NCT04797611 randomized controlled trial (RCT) period (day 113).
Time Frame: 3 months (NCT04797611 RCT: Day 29 - Day 113; this OLE: Day 113 to Day 197)
Population: This population received passive treatment during the RCT that preceded this OLE study during which they received active treatment. Only participants who completed the assessments at least once during the pre-treatment baseline period and at both the RCT end of treatment visit and the end of treatment period 1 visit during this OLE are included in the results posted. Full data collection was not completed as the study terminated prior to collection of outcome assessments for all participants.
Measure: Mean (95% Confidence Interval); unit: change in score on a scale from baseline
Arm/Group | Randomized Controlled Trial (RCT) Passive Treatment | Open Label Extension (OLE) Active Treatment
Number analyzed (Participants) | 50 | 50
change in score on a scale from baseline | -0.03 [-1.11 to 1.05] | 0.60 [-0.67 to 1.87]

3. Secondary Outcome: Change From Baseline in the Clinical Global Impression - Improvement (CGI-I)
Description: The CGI-I is a clinician assessment the extent of clinically meaningful change that has occurred in the patient's illness at day 197/365 relative to a baseline state (assessed at day 29). Changes in all aspects of Parkinson's disease (e.g., motor symptoms, non-motor symptoms and complications of anti-Parkinsonian medications) are considered. A "0" corresponds to no change, higher magnitude positive values correspond to greater improvements, and higher magnitude negative scores correspond to increased worsening. Scores range from -3 to +3 (-3 = very much worse, -2 = much worse, -1 = minimally worse, 0 = no change, 1=minimally improved, 2=much improved, 3=very much improved).
Time Frame: RCT: from Baseline (Day 29) up to 3 months (Day 113); OLE: from Baseline (Day 29) up to 11 months (Day 365)
Population: This population received passive treatment during the NCT04797611 RCT that preceded the active treatment received in this OLE study. Only participants who completed the assessments at least once during the RCT's pre-treatment baseline period, the RCT's end of treatment visit, and this OLE's end of treatment period 1 visit are included in the results posted. Full data collection was not completed as the study terminated prior to collection of outcome assessments for all participants.
Measure: Count of Participants; unit: Participants
Groups:
- Randomized Controlled Trial (RCT) Passive Treatment: This group received passive treatment with the study device in a randomized controlled trial that immediately preceded this open label extension during which participants received active (i.e., time-varying caloric vestibular simulation). Data is provided for change after the 12 weeks of passive treatment in the randomized controlled trial.
- Open Label Extension (OLE) Active Treatment: This group received passive treatment with the study device in a randomized controlled trial that immediately preceded this open label extension during which participants received active (i.e., time-varying caloric vestibular simulation). Data is provided for change after the 12 weeks of active treatment in the open label extension relative to the pre-treatment baseline in the randomized controlled trial.
Arm/Group | Randomized Controlled Trial (RCT) Passive Treatment | Open Label Extension (OLE) Active Treatment
Number analyzed (Participants) | 66 | 66
Participants
  1 - Very Much Improved | 0 | 0
  2 - Much Improved | 12 | 10
  3 - Minimally Improved | 22 | 23
  4 - No Change | 23 | 17
  5 - Minimally Worse | 7 | 11
  6 - Much Worse | 2 | 5
  7 - Very Much Worse | 0 | 0

4. Secondary Outcome: Change From Baseline in the International Parkinson and Movement Disorder Society Unified Parkinson's Disease Rating Scale Part III: Motor Examination (MDS-UPDRS Part III)
Description: The MDS-UPDRS Part III is a 33-item assessment of motor function evaluated by a trained blinded rater. Each item has five response options linked to accepted clinical terms (0/normal, 1/slight, 2/mild, 3/moderate, and 4/severe) for a total scoring range of 0-132. Higher scores indicate more severe motor symptoms. This secondary endpoint evaluates the change in MDS-UPDRS Part III score during the first treatment period of this open label extension (OLE) relative to the score at the end of the NCT04797611 randomized controlled trial (RCT) treatment period (day 113) for the passive-active treatment group compared to the change in MDS-UPDRS Part III score during the RCT treatment period relative to the pre-treatment baseline.
Time Frame: 3 months (NCT04797611 RCT: Day 29 - Day 113; this OLE: Day 113 to Day 197)
Population: This population received passive treatment during the RCT that preceded this phase of the study and active treatment in this OLE. Only participants who completed the assessments at least once during the RCT's pre-treatment baseline period and end of treatment visit and who completed the end of treatment period 1 visit during this OLE are included in the results posted. Full data collection was not completed as the study terminated prior to collection of outcome assessments for all participants.
Measure: Median (Inter-Quartile Range); unit: change in score on a scale from baseline
Arm/Group | Randomized Controlled Trial (RCT) Passive Treatment | Open Label Extension (OLE) Active Treatment
Number analyzed (Participants) | 58 | 58
change in score on a scale from baseline | 3.0 [-3.0 to 7.0] | -1.5 [-8.0 to 7.3]

5. Secondary Outcome: Change From Baseline in the Parkinson's Disease Quality of Life Questionnaire Summary Index (PDQ-39 SI)
Description: The PDQ-39 SI is a 39-item patient-reported quality of life measure that assesses how often people living with PD are affected across 8 dimensions of daily living covering: mobility (10 items), activities of daily living (6 items), emotional well-being (6 items), stigma (4 items), social support (3 items), cognition (4 items), communication (3 items), and bodily discomfort (3 items). Answers for each item range from 0/never to 4/always. Each dimension is scored by summing the scores of each item, dividing that maximum possible score of all items in the dimension, and then multiplying by 100. The total score (the SI score) is the sum of all dimension scores divided by 8 and ranges from 0-100, the higher the total score the greater the health problems).
  This endpoint compares the change in the PDQ-39 total score taken at the end of the RCT treatment period to the total score obtained during the OLE's first treatment period.
Time Frame: 3 months (NCT04797611 RCT: Day 29 - Day 113; this OLE: Day 113 to Day 197
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: change in score on a scale from baseline
Arm/Group | Randomized Controlled Trial (RCT) Passive Treatment | Open Label Extension (OLE) Active Treatment
Number analyzed (Participants) | 46 | 46
change in score on a scale from baseline | -2.20 [-6.93 to 12.10] | 0.15 [-2.68 to 2.60]

6. Secondary Outcome: Change From Baseline in the Combined Measure of The International Parkinson and Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS): Parts I, II and III
Description: The MDS-UPDRS evaluates motor (Parts I and III) and non-motor (Part II) experiences and complications of Parkinson's disease (PD) to characterizes the extent and burden of disease. Each question has five response options linked to accepted clinical terms: (0/normal, 1/slight, 2/mild, 3/moderate, and 4/severe)/evaluations and are divided across Part I (13 questions, 52 possible points), Part II (13 questions, 52 possible points), and Part III (33 questions based on 18 items, several with right, left or other body distribution scores, 132 possible points). The Combined Score is the sum of the points for all three Parts and ranges from 0 to 236. The higher the score, the more progressed (i.e., worse) is the disease state. The more negative the change score the greater the symptomatic improvement.
Time Frame: 3 months (NCT04797611 RCT: Day 29 - Day 113; this OLE: Day 113 to Day 197
Population: This population received passive treatment during the RCT that preceded this phase of the study and active treatment in this OLE. Only participants who completed the assessments at least once during the RCT's pre-treatment baseline period and the RCT's end of treatment visit and at the end of this OLE's treatment period 1 visit are included in the results posted. Full data collection was not completed as the study terminated prior to collection of outcome assessments for all participants.
Measure: Median (Inter-Quartile Range); unit: change in score on a scale from baseline
Arm/Group | Randomized Controlled Trial (RCT) Passive Treatment | Open Label Extension (OLE) Active Treatment
Number analyzed (Participants) | 38 | 38
change in score on a scale from baseline | -1.0 [-5.0 to 6.3] | -1.5 [-8.8 to 10.0]

7. Other Pre Specified Outcome: Change From Baseline in the Mini-Balance Evaluation Systems Test
Description: The Mini-BESTest is a 14-item test scored on a 3-level ordinal scale that assesses dynamic balance in terms of anticipatory postural adjustments, reactive postural control, sensory orientation, and dynamic gait. Answers to each of the 14 items range from 0/severe difficulty to 2/normal (no difficulty) for a total possible score ranging from 0 to 28 points. The lower the score the more difficulty was encountered. This measure will be evaluated as a safety outcome to assess whether device therapy negatively impacts balance or gait for participants with Parkinson's disease (day 197 score)
Time Frame: 8 months
Population: Full data collection was not completed as the study terminated prior to collection of outcome assessments for all participants.
Groups:
- Experimental Treatment 1: Study participants will self-administer ~19-minute treatments twice daily in the home setting using a non-invasive brainstem modulation device. The device has been deemed as a nonsignificant risk for studies in Parkinson's disease by the United States Food and Drug Administration.
Arm/Group | Experimental Treatment 1
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: Change From Baseline in the Montreal Cognitive Assessment
Description: The MoCA assesses cognition over 6 domains: Memory, Executive function, Attention, Language, Visuospatial, and Orientation. Points across all 6 domains are summed, and this sum equals the total score (min 0 - max 30). A higher total score indicates better cognitive function; a positive score for difference in points indicates improvement. A total score of 26-30 reflects normal cognition. Mild cognitive impairment is associated with a total score of 18-25. Total scores of 10 - 17 indicate moderate cognitive impairment; a total score less than 10 shows severe cognitive impairment.
  The change (difference) in the Montreal Cognitive Assessment (MoCA) total score taken at baseline and, again, at the end of treatment visit is reported. A positive change in scores indicates improvement; whereas, a negative change in scores between baseline and end of treatment indicates worsening. The more positive the change score, the greater the improvement.
Time Frame: 8 months
Population: as for outcome 7
Arm/Group | Experimental Treatment 1
Number analyzed (Participants) | 0

9. Other Pre Specified Outcome: Change From Baseline in the Oral Symbol Digit Modality Test (Oral SDMT)
Description: The oral SDMT assesses cognition that primarily evaluates processing speed and sustained attention. It involves a substitution task where the test taker pairs specific numbers with given geometric figures using a reference key. The oral version of the test allows responses to be given verbally, making it suitable for individuals with motor disabilities or speech disorders. It is scored based on the number of correct substitutions made. The scoring range for the oral version of the SDMT is from 0 to 110, where the score represents the number of correct substitutions made within 90 seconds and the maximum score is 110 points. A higher score indicates better performance, as it reflects a faster cognitive processing speed.
  The change/difference in scores between the baseline and end of study treatment are reported. A positive change in scores indicates improvement. A negative change in scores indicates worsening.
Time Frame: 8 months
Population: as for outcome 7
Arm/Group | Experimental Treatment 1
Number analyzed (Participants) | 0

10. Other Pre Specified Outcome: Change From Baseline in the Parkinson's Disease Sleep Scale (PDSS-2)
Description: The PDSS-2 is a patient-completed clinical rating scale that assesses the frequency of sleep disturbances over the past week. Each question is scored between 0 ("never") and 4 ("very often"), and a total score is calculated by summing a patient's responses to each of the 15 questions (minimum 0 to maximum 60). It has three domains: 1) motor problems at night, 2) PD symptoms at night, and 3) disturbed sleep. Total score ranges from 0 to 60, with the score of each domain ranging from 0 to 20. Higher scores represent more nighttime sleep-related problems. A positive change in scores indicates worsening. A negative change in scores indicates improvement.
Time Frame: 8 months
Population: as for outcome 7
Arm/Group | Experimental Treatment 1
Number analyzed (Participants) | 0

11. Other Pre Specified Outcome: Change From Baseline in Epworth Sleepiness Scale (ESS)
Description: The ESS is a questionnaire used to assess daytime sleepiness. The scale consists of eight questions where respondents rate their likelihood of falling asleep in various situations on a scale from 0 to 3, with 0 indicating no chance and 3 indicating a high likelihood. The total score ranges from 0 to 24. Results from 0 to 10 show average (normal) daytime sleepiness; a result under 10 may not be cause for concern or it could identify you have trouble sleeping (insomnia). A result from 11 to 24 indicates excessive (abnormal) daytime sleepiness (10-14 is mild, 15-17 is moderate, and 18 or higher is severe).
  A positive change in scores indicates worsening. A negative change in scores indicates improvement.
Time Frame: 8 months
Population: as for outcome 7
Arm/Group | Experimental Treatment 1
Number analyzed (Participants) | 0

12. Other Pre Specified Outcome: Change From Baseline in the Parkinson Anxiety Scale (PAS)
Description: he PAS is a 12-item observer or patient-rated scale designed to measure the severity of anxiety symptoms in patients with Parkinson's disease (PD). It includes three subscales that evaluate persistent anxiety (1-5), anxiety episodes (6-9), and avoidance behavior (10-12). Each item is scored on a 5-point Likert scale, where a score of "0" indicates "not" or "never," and a score of "4" indicates "severe" or "almost always." The total score for each subscale is calculated by summing the scores of the respective items. The maximum score for the entire scale is 48 points. A higher score indicates more severe anxiety symptoms.
Time Frame: 8 months
Population: as for outcome 7
Arm/Group | Experimental Treatment 1
Number analyzed (Participants) | 0

13. Other Pre Specified Outcome: Change From Baseline in the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) Scale
Description: The FACIT-Fatigue assesses fatigue-related symptoms and their impact on daily functioning. The scale includes a five-item symptom subscale and an eight-item impact subscale, totaling 13 items.
  For each item, level of fatigue is rated as 0 (Not at all) to 4 (Very much so). To score the FACIT-Fatigue, all items' ratings are summed to create a single fatigue score with a range from 0 to 52. Higher scores represent less fatigue, while lower scores indicate more fatigue.
Time Frame: 8 months
Population: as for outcome 7
Arm/Group | Experimental Treatment 1
Number analyzed (Participants) | 0

14. Other Pre Specified Outcome: Change From Baseline in the Geriatric Depression Scale-15 (GDS-15)
Description: The GDS-15 is a short, self-report questionnaire to identify depression in older adults. It consists of 15 items that assess mental health based on feelings over the past week. 1 point is given for any answer indicating depression; 0 is given for any answer not indicating depression. The total score is the sum of all items and points given and ranges from 0-15, with higher scores indicating more depression.
Time Frame: 8 months
Population: as for outcome 7
Arm/Group | Experimental Treatment 1
Number analyzed (Participants) | 0

15. Other Pre Specified Outcome: Change in the Movement Disorder Society Non-Motor Rating Scale (MDS-NMS) Non-Motor Fluctuations (NMF) Subscale Score
Description: The MDS-NMS NMF is a rater completed subscale that assesses the degree of change (0/no change to 4/large change) in non-motor symptoms in relation to the timing of anti-parkinsonian medications across 8 domains (depression, anxiety, thinking/cognitive abilities, bladder symptoms, restlessness, pain, fatigue, and excessive sweating). The degree of change provided for each of the 8 domains are summed. This sum is then multiplied by the time spent in non-motor "off" state (1/Rarely to 4/Majority of time) to obtain the MDS-NMS NMF Total Score.
  Total possible scores for this scale measure range from 0 to 334. The higher the total score, the more progressed (i.e., worse) is the disease state.
Time Frame: 8 months
Population: as for outcome 7
Arm/Group | Experimental Treatment 1
Number analyzed (Participants) | 0

16. Other Pre Specified Outcome: Change From Baseline in the Unified Parkinson's Disease Rating Scale (UPDRS IV) Part IV
Description: The UPDRS measures the severity and progression of Parkinson disease. Part IV assesses motor complications and is scored with yes and no ratings. Scores range: 0-24. Higher scores are worse; 4 and below is mild while 13 and above is severe.
Time Frame: 8 months
Population: as for outcome 7
Arm/Group | Experimental Treatment 1
Number analyzed (Participants) | 0

17. Other Pre Specified Outcome: Change From Baseline in the Zarit Burden Interview (ZBI)
Description: The ZBI is a 22-item questionnaire designed to measure the extent to which a caregiver perceives their level of burden because of caretaking. Each item on the interview is a statement which the caregiver is asked to endorse using a 5-point scale, ranging from 0 (Never) to 4 (Nearly Always). Total scores are obtained by summing all items endorsed. Scores are interpreted as follows: 0 to 21 indicates little or no burden, 21 to 40 indicates mild to moderate burden, 41 to 60 indicates moderate to severe burden, and 61 to 88 indicates severe burden.
Time Frame: 8 months
Population: as for outcome 7
Arm/Group | Experimental Treatment 1
Number analyzed (Participants) | 0

18. Other Pre Specified Outcome: Change From Baseline in the Patient Reported Outcome - Parkinson's Disease (PRO-PD)
Description: he PRO-PD is a self-rating, 32 item, visual analog scale (VAS) that assesses severity of PD symptoms. Each item evaluates a common PD symptom, covering both motor and non-motor symptoms, and is scored on a range from 0 ("no problem") to 100 ("extreme problem") points. The scores for all items are summed to obtain a total score that can range from 0 to 3200. Higher scores indicate more severe symptoms or greater impact on the patient's life.
Time Frame: 8 months
Population: as for outcome 7
Arm/Group | Experimental Treatment 1
Number analyzed (Participants) | 0

19. Other Pre Specified Outcome: Change From Baseline in The Modified Schwab and England Activities of Daily Living Scale
Description: This single-item clinical outcome scale assesses the functional status of individuals with Parkinson's Disease (PD). It evaluates their ability to perform daily activities, ranging from complete independence to complete dependence, with scores given in 10% increments from 100% (completely independent) to 0% (bedridden). The higher the score the more independent the participant is.
Time Frame: 8 months
Population: as for outcome 7
Arm/Group | Experimental Treatment 1
Number analyzed (Participants) | 0

20. Other Pre Specified Outcome: Change From Baseline in EncephaLogTM 3 Meter Timed Up and Go (TUG) Test
Description: Encephalog is an app through which the 3 Meter TUG Test can be run to evaluate the risk of falls in adults. The patient sits in with their back against the chair back. At "go," the patient rises from the chair, walks 3 meters at a comfortable/safe pace, turns, walks back to the chair, and sits. Timing begins at "go" and stops when reseated. The test measures in seconds. Scores indicate levels of mobility and fall risk; the higher the score (i.e., the longer it takes), the worse the functional mobility and greater the risk of falls: 10 seconds or less - normal mobility; 11-20 seconds - normal limits for frail/elderly/disabled patients; 20 seconds or more - need assistance, further examination and intervention; 30 seconds or more - significant mobility issue.)
Time Frame: 8 months
Population: as for outcome 7
Arm/Group | Experimental Treatment 1
Number analyzed (Participants) | 0

21. Other Pre Specified Outcome: Change From Baseline in EncephaLogTM Finger Tapping Test
Description: EncephaLog™ is a smartphone app through which the finger tapping test is conducted. The finger tapping test provides a quantitative measure of bradykinesia. A participant taps the phone as quickly as possible for 10 seconds with their index finger. Both left and right hand are tested. Scoring counts the number of finger taps in 10 seconds. The higher the score the more severe the symptoms.
Time Frame: 8 months
Population: as for outcome 7
Arm/Group | Experimental Treatment 1
Number analyzed (Participants) | 0

22. Other Pre Specified Outcome: Change From Baseline in EncephaLogTM 10m Timed Up and Go (10m TUG)
Description: EncephaLog™ is a smartphone app that measures gait and that provides indication of risk of falls in adults. The patient sits in the chair with his/her back against the chair back. On the command "go," the patient rises from the chair, walks 10 meters at a comfortable and safe pace, turns, walks back to the chair and sits down. Timing begins at the instruction "go" and stops when the patient is seated. Shorter times indicate less dysfunction.
  Scores of ten seconds or less indicate normal mobility. Scores between 11 and 20 seconds are within normal limits for frail elderly and disabled patients.
  Scores greater than 20 seconds suggest the person may need assistance outside and indicates further examination and intervention.
  Scores of 30 seconds or more suggest the person may be prone to falls.
Time Frame: 8 months
Population: as for outcome 7
Arm/Group | Experimental Treatment 1
Number analyzed (Participants) | 0

23. Other Pre Specified Outcome: Change From Baseline in Unified Parkinson's Disease Rating Scale Part I (UPDRS I)
Description: The UPDRS measures the severity and progression of Parkinson disease. Part I assesses Non-Motor Experiences of Daily Living in terms of mentation, behavior, and mood and is scored on a 0-4 rating scale. Total scores range from 0-16 with higher scores indicating more severe symptoms.
Time Frame: 8 months
Population: as for outcome 7
Arm/Group | Experimental Treatment 1
Number analyzed (Participants) | 0

24. Other Pre Specified Outcome: Change From Baseline in Hoehn & Yahr (H&Y)
Description: The Hoehn & Yahr scale is used to describe the progress of Parkinson's disease. Scoring is based on the level/stage of clinical disability described by severity of motor symptoms. Stage 1: Unilateral involvement only, usually with minimal or no functional disability. Stage 1.5: Unilateral and axial involvement. Stage 2: Bilateral involvement without impairment of balance. Stage 2.5: Mild bilateral disease with recovery on pull test. Stage 3: Bilateral disease with mild to moderate disability and impaired postural reflexes; physically independent. Stage 4: Severely disabling disease, still able to walk or stand unassisted. Stage 5: Confinement to bed or wheelchair unless aided. The greater the stage description, the more advanced the disease.
Time Frame: 8 months
Population: as for outcome 7
Arm/Group | Experimental Treatment 1
Number analyzed (Participants) | 0

25. Other Pre Specified Outcome: Change From Baseline in Patient Global Impression of Improvement
Description: a patient determined scale to assess how much their illness has improved or worsened relative to a baseline state at the beginning of the intervention.The Patient Global Impression of Improvement (PGI-I) is a tool used to measure a patient's perception of their condition following treatment. It is a single-item questionnaire that asks patients to rate their perceived change in condition on a scale from 1 (very much better) to 7 (very much worse).
Time Frame: 8 months
Population: as for outcome 7
Arm/Group | Experimental Treatment 1
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 8 months
Description: The clinicaltrials.gov definitions of AE and SAE were used
Groups:
- Experimental: Passive-active: This group received passive treatment with the study device in a randomized controlled trial that immediately preceded this open label extension trial during which participants received active (i.e., time-varying caloric vestibular stimulation) treatment.
  Treatment was ~20 minutes, 2x per day for 12 weeks, then a follow-up period without treatment for 16 weeks, then another 8 week treatment period with the active treatment.
- Experimental: Active-active: This group received active (i.e. time-varying caloric vestibular stimulation) treatment with the study device in a randomized controlled trial that immediately preceded this open label extension trial during which participants received active treatment. Data obtained from this group was only utilized for exploratory outcome measures.
  Treatment was ~20 minutes, 2x per day for 12 weeks, then a follow-up period without treatment for 16 weeks, then another 8 week treatment period with the active treatment.
Arm/Group | Experimental: Passive-active | Experimental: Active-active
All-Cause Mortality (participants affected / at risk) | 1/69 | 1/79
Serious Adverse Events (participants affected / at risk) | 7/69 | 6/79
Other Adverse Events (participants affected / at risk) | 51/69 | 42/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Passive-active (N=69) | Experimental: Active-active (N=79)
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bilateral Pleural Effusions (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cerebral Vascular Accident (Nervous system disorders) | 1 (1) | 0 (0)
Right Knee Replacement surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Multiple Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Partial Small Bowl Obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute Gastroenteritis with Dehydration (Gastrointestinal disorders) | 0 (0) | 1 (1)
ESCHERICHIA COLI URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Weakness secondary to urosepsis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Passive-active (N=69) | Experimental: Active-active (N=79)
COVID-19 (Infections and infestations) | 9 (9) | 12 (12)
Fall (Injury, poisoning and procedural complications) | 16 (24) | 12 (25) — secondary to a trip, gait freezing, imbalance/slipping, or orthostatic hypotension
Dizziness (Nervous system disorders) | 9 (11) | 5 (7) — An episode of lightheadedness, dizziness, or worsening dizziness
Nasopharyngitis (Infections and infestations) | 6 (7) | 7 (8) — cold, head cold, common cold, etc.
Medical device site discomfort (General disorders) | 6 (6) | 2 (2)
Nausea (Gastrointestinal disorders) | 5 (6) | 4 (4) — An incident of nausea

LIMITATIONS AND CAVEATS:
This study was terminated early due to lack of device effectiveness demonstrated in STEM-PD RCT (NCT04797611) prior to final outcome measures being collected for all participants enrolled in this OLE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-05-10): https://cdn.clinicaltrials.gov/large-docs/18/NCT04799418/Prot_000.pdf
  • Statistical Analysis Plan (2025-04-22): https://cdn.clinicaltrials.gov/large-docs/18/NCT04799418/SAP_002.pdf